CLINICAL TRIAL: NCT05882916
Title: Reaching the Last 20%: a Targeted HIV Self-test Secondary Distribution Intervention to Engage High-risk Men in Kenya
Brief Title: Reaching the Last 20% (the Pamoja Kwa Afya Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sue Napierala (Other)
Collaborators: Impact Research & Development Organization (Other); University of Pennsylvania (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Sue Napierala, Principle Investigator, RTI International
Organization: RTI International (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0218622
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: Self-testing; Secondary distribution; Men who purchase sex; Women who sell sex; HIV

STUDY DESIGN:
Intervention Model Description: randomized stepped wedge trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIV self-test secondary distribution (Experimental): The investigators will provide women who sell sex enrolled in the study with multiple World Health Organization (WHO) and Kenya-approved oral fluid-based HIV self-test kits. Participants will be counseled to secondarily distribute self-tests to their male transactional sex partners. Self-test kits will contain instructions for use and tailored information on clinic locations and hours within the cluster, the benefits of early ART use, and the availability and benefits of PrEP.
  Interventions: Device: HIV self-testing; Behavioral: Behavioral economic 'nudges'

INTERVENTIONS:
Device: HIV self-testing — Oral fluid-based HIV self-test kits for secondary distribution
Behavioral: Behavioral economic 'nudges' — Salient information for men included with the self-test kit on clinic location and hours within their cluster, and pilot-tested messaging on the importance of early ART initiation, and the availability and benefits of PrEP

SUMMARY:
This cluster randomized controlled trial will test whether the provision of multiple oral fluid-based HIV self-test kits to women who sell sex (WSS) to secondarily distribute to their male partners who purchase sex can promote uptake of HIV service use by male partners. The study will recruit adult women who report exchanging sex for compensation in Kisumu and Siaya counties in Western Kenya. In clusters randomized to the intervention, WSS will be given multiple HIV self-tests and counseled to distribute them to men who purchase sex (MPS). Self-test kits will contain instructions for use and tailored information on clinic location and hours within the cluster, and pilot-tested messaging on the benefits of antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP). In control clusters, standard of care HIV services will continue to be available. To objectively assess impacts of the intervention on post-HIVST linkage outcomes, the investigators will monitor use of HIV services by men at HIV clinics in both study arms on a monthly basis. Our goal will be to determine whether confirmatory testing (primary outcome), case diagnoses, ART initiation, and PrEP initiation by men in intervention clusters are higher than in control clusters. Mixed methods research will be utilized to conduct a process evaluation to assess mechanisms that may have impacted intervention effectiveness, pathways for linkage among MPS, and support for men's linkage to HIV services under a secondary distribution model. Cost-effectiveness analyses will also be undertaken.

DETAILED DESCRIPTION:
Limited use of HIV services by those at highest risk is one of the primary reasons for continued HIV transmission in sub-Saharan Africa. Identifying and engaging these individuals-particularly the 20% of people living with HIV who are unaware of their status-is a major challenge that is not being met by existing service delivery approaches. Men who purchase sex (MPS) are of particularly high priority because they are twice as likely to be HIV-infected as other men and are inherently challenging to identify and reach with HIV services. The proposed project will take place in the region of Kenya with the highest HIV prevalence and seeks to promote engagement in HIV testing, prevention, and care by MPS. Preliminary data demonstrate that "secondary distribution" of HIV self-tests by women who sell sex (WSS) to their sexual partners is acceptable, feasible, and safe and leads to high male partner testing. However, the use of post-self-test services has seldom been promoted or measured in a secondary distribution model. Our interdisciplinary and experienced team of Investigators will address this key gap.

This project will use a stepped wedge trial design to test an innovative, well-targeted HIV self-test secondary distribution intervention to promote uptake of HIV services by MPS. Clusters served by Ministry of Health-supported HIV clinics will be randomized to the start time to receive the secondary distribution intervention. The investigators will recruit WSS from key population clinics and transactional sex "hot spots." WSS will be provided with oral fluid-based HIV self-tests and encouraged to distribute them to their male transactional sex partners. Self-test kits will include salient information for men on clinic location and hours within their cluster, and pilot-tested messaging on the importance of early ART initiation, and the availability and benefits of PrEP. In Aim 1, the investigators will evaluate programmatic data from HIV clinics in study clusters to objectively determine the intervention's impact on uptake of confirmatory testing, HIV case diagnoses, and ART initiation and PrEP initiation by men. In Aim 2, the investigators will conduct a process evaluation to characterize factors influencing intervention effectiveness. The investigators will assess secondary distribution patterns and characterize the MPS population receiving self-tests through quantitative program data and a follow-up questionnaire among enrolled WSS. The investigators will use qualitative data obtained through in-depth interviews with MPS, WSS and clinic staff to explore pathways and contextual factors influencing whether men accessed post-test services. In Aim 3, the investigators will compute the incremental cost-effectiveness of our intervention to inform decisions about broader implementation. This project has the potential to break new ground on ways to engage high-risk and hard-to-reach populations in HIV services. If effective, our approach could be readily adapted to other settings and help advance global goals for HIV elimination.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥18 years
* Reports exchanging sex for compensation with ≥2 men in the past month
* Engages in sex for compensation in the intervention cluster catchment area
* Willing to participate in a brief questionnaire 6 weeks after enrollment
* Plan to remain in the area of study recruitment for the next 8 weeks

Exclusion Criteria:

* Unwilling or unable to provide informed consent for participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as female
Enrollment: 5000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
HIV testing | 3 months
  The count of adult men from each cluster who completed an HIV test at the clinic within the intervention versus control period.

SECONDARY OUTCOMES:
HIV case diagnoses | 3 months
  The test positivity rate at the clinic (proportion of men who obtain an HIV-positive result) within the intervention versus control period.
ART and PrEP initiation | 3 months
  The count of adult men from each cluster who initiated ART or PrEP at the clinic within the intervention versus control period.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Napierala, PhD, MPH, Principal Investigator — RTI International
Locations (1):
- Impact Research and Development Organization (IRDO), Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thirumurthy H, Masters SH, Mavedzenge SN, Maman S, Omanga E, Agot K. Promoting male partner HIV testing and safer sexual decision making through secondary distribution of self-tests by HIV-negative female sex workers and women receiving antenatal and post-partum care in Kenya: a cohort study. Lancet HIV. 2016 Jun;3(6):e266-74. doi: 10.1016/S2352-3018(16)00041-2. Epub 2016 Apr 8. PMID 27240789
- [Background] Lynch M, Pentecost BL, Littler WA, Stockley RA. The distribution of antibodies to streptokinase. Postgrad Med J. 1996 May;72(847):290-2. doi: 10.1136/pgmj.72.847.290. PMID 8761502
- [Background] Napierala S, Bair EF, Marcus N, Ochwal P, Maman S, Agot K, Thirumurthy H. Male partner testing and sexual behaviour following provision of multiple HIV self-tests to Kenyan women at higher risk of HIV infection in a cluster randomized trial. J Int AIDS Soc. 2020 Jun;23 Suppl 2(Suppl 2):e25515. doi: 10.1002/jia2.25515. PMID 32589354
- [Background] Masters SH, Agot K, Obonyo B, Napierala Mavedzenge S, Maman S, Thirumurthy H. Promoting Partner Testing and Couples Testing through Secondary Distribution of HIV Self-Tests: A Randomized Clinical Trial. PLoS Med. 2016 Nov 8;13(11):e1002166. doi: 10.1371/journal.pmed.1002166. eCollection 2016 Nov. PMID 27824882